CLINICAL TRIAL: NCT06532656
Title: A Phase 2/3, Open-Label Study to Evaluate the Pharmacokinetics, Safety, and Antiviral Activity of Bictegravir/Lenacapavir in Children and Adolescents With HIV-1
Brief Title: Study of Bictegravir/Lenacapavir in Children and Adolescents With HIV-1
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-621-6463; 2023-509428-16 (Other: European Medicines Agency)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Participants Aged ≥ 12 to < 18 years with Weight ≥ 35 kg: BIC/LEN 75/50 mg FDC (Experimental): Participants will receive a 2-day oral loading dose of LEN (600 mg) on Days 1 and 2 and daily oral BIC/LEN 75/50 mg starting on Day 1 through Week 48.
  Following Week 48, participants will have an option to continue BIC/LEN in the extension period.
  Interventions: Drug: Lenacapavir; Drug: BIC/LEN FDC
- Cohort 2: Participants Aged ≥ 6 to < 12 years with Weight ≥ 25 kg to < 35 kg (Experimental): All participants will receive a 2-day oral loading dose of LEN, and daily oral BIC and LEN dose starting on Day 1 through Week 48. Dose in cohort 2 to be defined.
  Following Week 48, participants will have an option to continue BIC/LEN in the extension period.
  Interventions: Drug: Lenacapavir; Drug: BIC/LEN FDC
- Cohort 3: Participants Aged ≥ 2 to < 6 years with Weight ≥ 10 kg to < 25 kg (Experimental): All participants will receive a 2-day oral loading dose of LEN, and daily oral BIC and LEN dose starting on Day 1 through Week 48. Dose in cohort 3 to be defined.
  Following Week 48, participants will have an option to continue BIC/LEN in the extension period.
  Interventions: Drug: Lenacapavir; Drug: BIC/LEN FDC

INTERVENTIONS:
Drug: Lenacapavir — Tablets administered orally without regard to food
  Other Names: GS-6207
Drug: BIC/LEN FDC — Tablets administered orally without regard to food

SUMMARY:
The goal of this clinical study is to learn about the safety and tolerability of bictegravir/lenacapavir (BIC/LEN) and to learn how the study drug interacts with the body in virologically suppressed (VS) children and adolescents with human immunodeficiency virus type 1 (HIV-1) on a stable and complex antiretroviral (ARV) regimen. The study will also assess the safe loading dose of LEN and pharmacokinetics (PK) of BIC/LEN.

The primary objectives of this study are:

* To evaluate the steady-state PK of BIC and LEN and confirm the dose of the LEN loading dose and BIC/LEN FDC in VS children and adolescents with HIV-1.
* To evaluate the safety and tolerability of BIC/LEN through Week 24 in VS children and adolescents with HIV-1.

ELIGIBILITY:
Key Inclusion Criteria:

* Age and body weight at screening:

  * Cohort 1: ≥ 12 years to < 18 years weighing ≥ 35 kg.
  * Cohort 2: ≥ 6 years to < 12 years weighing ≥ 25 kg to < 35 kg.
  * Cohort 3: ≥ 2 years to < 6 years weighing ≥ 10 kg to < 25 kg.
* On a complex ARV regimen. Complex regimens are any ARV therapy that is not a single-tablet regimen taken once daily (eg, > 1 tablet or any other formulation a day).
* Documented plasma HIV-1 ribonucleic acid (RNA) levels must be < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is < 50 copies/mL) in the last 6 months prior to screening (at least 1 measure prior to screening).
* Plasma HIV-1 RNA levels < 50 copies/mL at screening.
* No documented or suspected resistance to integrase strand transfer inhibitors (mutations T66A/I/K, E92G/Q/V, G118R, F121C/Y, G140R, Y143C/H/R, S147G, Q148H/K/R, N155H/S, or R263K in the integrase gene).
* The following laboratory parameters at screening:

  * Estimated glomerular filtration rate ≥ 30 mL/min/1.73 m2 using the Bedside Schwartz formula.
  * Absolute neutrophil count > 0.50 cells/L (> 500 cells/mm3).
  * Hemoglobin ≥ 85 g/L (> 8.5 g/dL).
  * Platelets ≥ 50 cells/L (≥ 50,000 cells/mm3).
  * Hepatic transaminases (aspartate aminotransferase and alanine aminotransferase)

    ≤ 5 x upper limit of normal.
  * Total bilirubin ≤ 23 μmol/L (≤ 1.5 mg/dL) and direct bilirubin ≤ 7 μmol/L (≤ 0.4 mg/dL).

Key Exclusion Criteria:

* CD4 cell count < 200 cells/mm^3.
* CD4 percentage < 20%.
* Life expectancy ≤ 1 year.
* An opportunistic illness indicative of Stage 3 HIV diagnosed within the 30 days prior to screening.
* Evidence of active pulmonary or extrapulmonary tuberculosis within 3 months prior to screening.
* Acute hepatitis within 30 days prior to screening.
* Positive hepatitis C virus (HCV) antibody with detectable HCV RNA (participants positive for HCV antibody will have an HCV RNA test performed).
* Positive hepatitis B surface antigen (HBsAg) or positive hepatitis B virus (HBV) core antibody (antibody against hepatitis B core antigen [anti-HBc]) at screening. If a participant is negative for HBsAg and positive for anti-HBc but HBV DNA is undetectable, the participant may be enrolled.
* A history of or current decompensated liver cirrhosis (eg, ascites, encephalopathy, or variceal bleeding).Current alcohol or substance use judged by the investigator to potentially interfere with the participant's study compliance.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
PK Parameter: Cmax of BIC and LEN at Steady State | Day 1 up to Week 24, as appropriate
  Cmax is defined as the maximum observed concentration of drug at steady state.
PK Parameter: AUCtau of BIC and LEN at Steady State | Day 1 up to Week 24, as appropriate
  AUCtau is defined as the area under the concentration versus time curve over the dosing interval at steady state.
PK Parameter: Ctrough of BIC and LEN at Steady State | Day 1 up to Week 24, as appropriate
  Ctrough is defined as the observed drug concentration at the end of the dosing interval at steady state.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) Through Week 24 | First dose date up to Week 24
Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Through Week 24 | First dose date up to Week 24

SECONDARY OUTCOMES:
PK Parameter: AUClast for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  AUClast is defined as the area under the concentration versus time curve from time zero to the last quantifiable concentration at steady state.
PK Parameter: Tmax for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  Tmax is defined as the time (observed time point) of Cmax at steady state.
PK Parameter: Tlast for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  Tlast is defined as the time (observed time point) of Clast at steady state. Clast is defined as the last measurable concentration (above the quantification limit).
PK Parameter: T1/2 for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  T1/2 is defined as the terminal elimination half-life at steady state.
PK Parameter: CL for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  Clearance (CL) is the volume of plasma cleared of drug over a specified time period, at a steady state.
PK Parameter: Vz for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  Volume of distribution (Vz) is defined as the extent to in which the drug is distributed in the body tissue, rather than the plasma, to produce the desired effects at a steady state.
PK Parameter: λz for BIC and LEN at Steady State | Day 1 up to Week 48, as appropriate
  λz is defined as the terminal elimination rate constant, which determines the rate at which the drug will be eliminated from the body after it is absorbed and distributed at a steady state.
Percentage of Participants Experiencing TEAEs Through Week 48 | First dose date up to Week 48
Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities Through Week 48 | First does date up to Week 48
Proportion of Participants With Plasma HIV-1 RNA < 50 copies/mL and ≥ 50 copies/mL at Week 24 Based on the United States (US) Food and Drug Administration (FDA)-Defined Snapshot Algorithm | Week 24
Proportion of Participants With Plasma HIV-1 RNA < 50 copies/mL and ≥ 50 copies/mL at Week 48 Based on the United States FDA-Defined Snapshot Algorithm | Week 48
Change from Baseline in Clusters of Differentiation 4 (CD4) Cell Counts at Week 24 | Baseline, Week 24
Change from Baseline in CD4 Percentage at Week 24 | Baseline, Week 24
Change from Baseline in CD4 Cell Counts at Week 48 | Baseline, Week 48
Change from Baseline in CD4 Percentage at Week 48 | Baseline, Week 48
Acceptability and Palatability Summary of LEN Oral Loading Dose at Day 1 Assessed by Questionnaire | Day 1
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.
Acceptability and Palatability Summary of LEN Oral Loading Dose at Day 2 Assessed by Questionnaire | Day 2
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.
Acceptability and Palatability Summary of Oral BIC/LEN Fixed Dose Combination (FDC) at Day 1 Assessed by Questionnaire | Day 1
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.
Acceptability and Palatability Summary of Oral BIC/LEN FDC at Week 4 Assessed by Questionnaire | Week 4
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.
Acceptability and Palatability Summary of Oral BIC/LEN FDC at Week 24 Assessed by Questionnaire | Week 24
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.
Acceptability and Palatability Summary of Oral BIC/LEN FDC at Week 48 Assessed by Questionnaire | Week 48
  Palatability and acceptability assessed by a numeric response between numbers 1-5. Higher scores indicate better palatability and acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (21):
- United States (4):
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Grady Ponce de Leon Center, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
- Helios Salud S.A, Buenos Aires, Argentina
- Italy (2):
  - ASST FBF Sacco Ospedale Sacco, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesu, UOS Infezioni Complesse e Perinatali, Roma
- South Africa (11):
  - FAMCRU Ukwanda School for Rural Health, Cape Town
  - Be Part Yoluntu, Cape Town
  - Durban International Clinical Research Site, Enhancing Care Foundation, Durban
  - Monti Clinical Research Centre, East London
  - Perinatal HIV Research Unit, Johannesburg
  - Wits RHI Shandukani Research Centre CRS, Johannesburg
  - Nkanyezi VIDA Research Unit, Johannesburg
  - Khomanani Health Research and Wellness Centre, Ka-Majosi
  - Clinical Research Institute of South Africa (CRISA), KwaDukuza
  - The Aurum Institute: Pretoria Clinical Research Centre, Pretoria
  - Setshaba Research Centre, Soshanguve
- Spain (3):
  - Hospital General Universitario Gregorio Marano, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06532656